CLINICAL TRIAL: NCT05551156
Title: The Role of Therapy Dogs in Reducing Depression, Anxiety, and Loneliness Among Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Purina Mills, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20023539
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Hospitalized Children

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal-assisted interaction (Experimental): A dog-handler team will visit participants in their hospital room
  Interventions: Behavioral: Animal-assisted interaction
- Conversational interaction (Experimental): Conversational interaction with the participants and the dog-handler
  Interventions: Behavioral: Conversational interaction
- Treatment as usual (No Intervention): Participants will received the regular services currently being received in the hospital

INTERVENTIONS:
Behavioral: Animal-assisted interaction — Visits will occur on 3 consecutive days during your participant's inpatient hospital stay. A dog-handler team or a handler alone will visit participants with a dog for approximately 20 minutes at a convenient time for the participant. During this visit, the participant will be able to pet the dog if they wish. The handler will talk with the participants about the dog, the weather, sports, or other light topics. Participants can also suggest light topics to talk about as well.
  Arms: Animal-assisted interaction
Behavioral: Conversational interaction — Visits will occur on 3 consecutive days during your participant's inpatient hospital stay. A dog-handler team or a handler alone will visit participants without a dog for approximately 20 minutes at a convenient time for the participant. During this visit, the handler will talk with the participants about the weather, sports, or other light topics. Participants can also suggest light topics to talk about as well.
  Arms: Conversational interaction

SUMMARY:
The purpose of this research study is to test whether an animal-assisted intervention (AAI) is better than conversation with another person or treatment as usual for improving mood, anxiety, loneliness, quality of life, and indicators of health care services such as number of hospitalizations, length of hospital stay, and cost of services for children and adolescents.

DETAILED DESCRIPTION:
Rationale: Loneliness is linked to a number of health threats, is considered to be as harmful as smoking 15 cigarettes a day, and is potentially more dangerous than obesity. Loneliness was considered to be at epidemic proportions prior to the COVID-19 pandemic. The resulting need for social distancing has exacerbated loneliness and other mental health concerns. Loneliness is associated with significant morbidity and mortality risks among people with Mental Illness (MI). As many as 70% of community-dwelling adults with MI endorse experiencing loneliness, which increases exponentially with the number of co-morbid psychiatric diagnoses. A growing body of evidence indicates that companion animals offer a number of health and wellbeing benefits. Interacting with a trained therapy animal as part of an animal-assisted interaction (AAI) may provide social support for patients with mental illness, thus reducing the risk of loneliness. The use of AAIs for hospitalized patients with MI as a strategy for reducing loneliness has been understudied. Scientists and practitioners need clear answers to some key questions before specific recommendations can be made.

Hypothesis/Objectives: 1. Evaluate the feasibility of a therapy dog visitation intervention (AAI) over four consecutive days on an inpatient psychiatry unit, compared to a conversational control intervention (CC), and a treatment as usual control condition (TU) in psychiatric inpatients; 2. Assess the efficacy of an AAI over four consecutive days, compared to CC, and a treatment as usual control condition (TU) in psychiatric inpatients; 3. Obtain information required to estimate sample size for a large randomized controlled trial (RCT) of a therapy dog visitation program in the population of psychiatric inpatients, combined with already funded pilot data from a sample of older adults to calculate power, determine sample size, and pursue federal funding for a large scale, multi-site, clinical trial.

Study Design and Methods: The proposed study employs a three-group RCT design to examine study implementation feasibility and effects of AAI compared to CC and TU conditions. The investigators will randomize 60 psychiatry inpatients to one of three conditions (AAI, CC, or TU) for a four-day treatment period.

Preliminary Data: Demonstrated reductions in anxiety and fear in hospitalized psychiatric patients following brief AAI provide a foundation for this work.

Expected Results: The investigators anticipate that patients will demonstrate greater improvements in the primary outcome of loneliness, and in the secondary mental health and well-being outcomes of anxiety, depression, HRQOL and mood in the therapy dog visitation program compared to the CC and TU conditions from phase 1-4 and from pre to post intervention during phase 2. The investigators anticipate that at least 50% of patients approached will consent to participation in the study. The investigators anticipate greater than 75% adherence (session completion) and less than 25% attrition (failure to attend sessions) in the AAI and CC groups. The investigators anticipate similar rates of completion in phase 3 and phase 4 assessments in the three groups, with greater failure longer after study completion. The investigators anticipate that a high proportion (at least 75%) of patients will report satisfaction with the AAI (phase 3) and that the proportion will be higher than for the CC. The investigators will explore differences in willingness to consent, instrument completion (rates of missing data), and adherence and attrition across conditions.

Potential Impact on Human-Animal Bond Research: This proposal uniquely addresses loneliness, a critical mechanism that contributes to mortality and potential morbidity among people with serious mental illness. Completing the proposed research will allow us to collect necessary pilot data to support a larger, funded, fully powered RCT to test the effectiveness of therapy dog visitation as an adjunctive treatment for people with serious mental disorders . If findings support the superior efficacy of therapy dog visitation compared to other conditions, this information can be used not only to support its use as an inpatient intervention, but to provide a foundation for studying its utility in community-based mental health contexts, such as assertive community treatment, wellness action and recovery programs, and in supportive housing.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for children:

* Projected to be admitted to the hospital for the upcoming five days
* between 8-17 years of age
* speak English
* be able to provide assent (understand what the study is about and what activities are involved)

Inclusion criteria for parents:

* Age 18+
* English-speaking
* Access to working phone, email, or address so that follow-up measures can be completed/sent.

Exclusion Criteria:

Exclusion criteria for children:

* Fear of or allergy to dogs
* documented contact precautions
* cognitive impairment that prevents consent/assent or completion of measures
* inability to participate in the study in the clinical judgment of their healthcare provider.

Exclusion criteria for parents:

* Inability to understand documents written in English
* Fear of or allergy to dogs

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Change in Depression | Baseline to end of treatment (about 5 days), 1 month after treatment
  Depressive symptomology will be measured with the 13-item Mood and Feelings Questionnaire (MFQ) which are rated on a 3 point scale. Higher scores indicate greater depression.
Change in Anxiety | Baseline to end of treatment (about 5 days), 1 month after treatment
  Anxiety will be measured using the 6-item state scale of the State-Trait Anxiety Inventory for Children (STAI-C) which are rated on a 3 point scale. Higher scores indicate more anxiety.
Change in Mood | Baseline to end of treatment (about 5 days), 1 month after treatment
  Mood will be measured using the Smiley Face Assessment Scale in which participants select which face fits their current mood. The scale depicts five emoticons from very sad to very happy.
Change in Loneliness | Baseline to end of treatment (about 5 days), 1 month after treatment
  Child loneliness will be assessed using the 11-item version of the De Jong Gierveld Loneliness Scale for children which are answered on a 5 point scale. Higher scores indicate greater loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Gee, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Administration HRaS. The Loneliness Epidemic. https://www.hrsa.gov/enews/past-issues/2019/january-17/loneliness-epidemic. Published 2019. Accessed January 23, 2021.
- [Background] Dell NA, Pelham M, Murphy AM. Loneliness and depressive symptoms in middle aged and older adults experiencing serious mental illness. Psychiatr Rehabil J. 2019 Jun;42(2):113-120. doi: 10.1037/prj0000347. Epub 2019 Jan 21. PMID 30667243
- [Background] Meltzer H, Bebbington P, Dennis MS, Jenkins R, McManus S, Brugha TS. Feelings of loneliness among adults with mental disorder. Soc Psychiatry Psychiatr Epidemiol. 2013 Jan;48(1):5-13. doi: 10.1007/s00127-012-0515-8. Epub 2012 May 9. PMID 22570258
- [Background] Wells DL. The state of research on human-animal relations: implications for human health. Anthrozoös. 2019;32(2):169-181.
- [Background] Krause-Parello CA, Gulick, E.E., Basin, B. Loneliness, depression, and physical activity in older adults: The therapeutic role of human-animal interactions. Anthrozoös. 2019;32(2):239-254.
- [Background] Barker SB, Dawson KS. The effects of animal-assisted therapy on anxiety ratings of hospitalized psychiatric patients. Psychiatr Serv. 1998 Jun;49(6):797-801. doi: 10.1176/ps.49.6.797. PMID 9634160
- [Background] Barker SB, Pandurangi AK, Best AM. Effects of animal-assisted therapy on patients' anxiety, fear, and depression before ECT. J ECT. 2003 Mar;19(1):38-44. doi: 10.1097/00124509-200303000-00008. PMID 12621276